CLINICAL TRIAL: NCT03437980
Title: Can Propofol Procedural Sedation Implementation Increase the Acceptance of Spinal Anesthesia During Cesarean Section?
Brief Title: Propofol Spinal Procedural Sedation for Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Alaa Mazy Mazy, associate professor of anesthesia and surgical intensive care, Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: R.18.02.23
Record Dates: First submitted 2018-02-04; First posted 2018-02-19 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Patient Compliance
MeSH Terms: conditions — Patient Compliance | interventions — Propofol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- propofol spinal acceptance (Experimental): The surgeon and the anesthetist will discuss the exclusion criteria. Then they will discuss the information's about spinal and general anesthesia with the illegible patients, also reply the patient's questions in a preoperative visit. The primary decision for the patient; either spinal or general anesthesia will be recorded.
  The patients refusing spinal anesthesia will be discussed again to detect the rate of acceptance of spinal anesthesia if propofol sedation is ensured during the procedure to provide a painless spinal injection. The final decision will be applied; either spinal with procedural sedation, or general anesthesia.
  Interventions: Drug: propofol

INTERVENTIONS:
Drug: propofol — A bolus of 0.7 mg/kg will be given initially, additional incremental doses of 20 mg propofol will be given if the patient complained of pain or moved arms towards the back. Patients will be sitting on the middle of the operating table facing towards the table's foot. The table's foot will be dropped 45 degrees for a comfortable chair position, Monitoring through pulse oximeter (SaO2), non-invasive blood pressure (NIBP) adjusted every 2 minutes automatic measuring and capnography tube in contact with nostrils.
  Other Names: propofol procedural sedation

SUMMARY:
Patient's safety and satisfaction are major concerns of anesthesiologists and obstetricians. According to evidence, guidelines and quality markers, regional anesthesia is preferred over general anesthesia in obstetric surgery. A high level of anxiety is present in obstetric patients preoperatively. Patients with high anxiety tend to prefer general anesthesia for cesarean section. The anxiety can be reduced variably by non-pharmacologic and pharmacologic methods. The evidence supports the benefits of procedural sedation for distressed, anxious pregnant women.

DETAILED DESCRIPTION:
Propofol provides short onset, rapid predictable action, anxiolysis and amnesia and it is more effective than benzodiazepines. Using propofol infusion in low doses during spinal injection in CS did not adversely affect the Apgar scores or the neurological and adaptive fetal outcomes. The general consensus is that procedural sedation is not a routine for spinal interventions, but required for anxious patients. Our hypothesis is that, with the high prevalence of maternal anxiety during cesarean section, ensuring painless comfortable spinal anesthesia may increase the acceptance rate of regional anesthesia during cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective cesarean section,
* Age: 18 - 40 years,
* American Society of Anesthesiologists I - III,
* Patients may present any of the following conditions:
* Respiratory diseases as bronchial asthma
* Hepatic compromise,
* Preeclampsia,
* Anemia with hemoglobin 10 g/dl,
* Previous sections,
* Obese with BMI more than 35%,
* Any criteria of difficult intubation, Compromised fetus as premature delivery, History of complications or non-satisfaction after general anesthesia during previous cesarean section,

Exclusion Criteria:

* Patients refusing to participate in the study,
* Known psychiatric disease,
* Addiction medications,
* Communication barrier,
* Absolute or relative contraindication for spinal anesthesia,
* Bad obstetric history, complicated pregnancy, congenital fetal anomaly.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — patients scheduled for an elective cesarean section.
Enrollment: 228 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-07-10 (Actual); Study Completion 2018-09-10 (Actual)

PRIMARY OUTCOMES:
The rate of acceptance of spinal anesthesia if propofol sedation is added during the procedure. | 30 minutes preoperative.
  percent

SECONDARY OUTCOMES:
The rate of initial acceptance of spinal anesthesia without sedation. | 30 minutes preoperative.
  percent
The anxiety score. | 30 minutes preoperative,10 minutes after spinal injection, and 30 minutes after stay at recovery room.
  by the visual analogue score from 0-10, where 10 is the maximum anxiety level.

OTHER OUTCOMES:
The patient satisfaction regards the spinal anesthesia decision. | 30 minutes at recovery room.
  The patients express thier satisfaction with the spinal decision on a visual analogue score, ranging from 0 to 10, where 0 is the minimum and 10 is the maximum satisfaction level.
The total utilized dose of propofol. | 1 minute after completion of spinal procedure, and 5 minutes at the end of cesarean section.
  milligram
The rate of premature termination of spinal procedure (failure rate). | 20 minutes preoperative.
  percent
The sedation score. | determined 1 minutes after following spinal injection. then again after 10 minutes.
  using modified Ramsay scale, 1. Anxious, 2. Cooperative, oriented, tranquil. 3. Responsive to commands only. If Asleep. 4. Brisk response to light glabellar tap or loud auditory stimulus. 5. Sluggish response to light glabellar tap or loud auditory stimulus.
The infant Apgar score. | 0 and 5 minutes after delivery.
  A measure of the physical condition of a newborn infant. Adding points (2, 1, or 0) for heart rate, respiratory effort, muscle tone, response to stimulation, and skin coloration; ranges from 0- 10, score of ten represents the best possible condition.
Patient's choice of anesthesia next time. | 30 minutes after shifting the patient to recovery room.
  spinal or general anesthesia.
The incidence of desaturation during propofol spinal procedural sedation. | 20 minutes preoperative.
  in percent, desaturation defined as oxygen saturation less than 90%
The incidence of hypotension during propofol spinal procedural sedation. | 20 minutes preoperative.
  in percent, hypotension defined as mean blood pressure less than 60 millimeter mercury.

CONTACTS AND LOCATIONS:
Locations (3):
- Egypt (3):
  - Delta Hospital, Al Mansurah, Dakahlya
  - Mansoura University Hospital, Al Mansurah, Dakahlya
  - Zagazig University Hospital, Zagazig, Sharkya

IPD SHARING:
Plan to Share IPD: Undecided